CLINICAL TRIAL: NCT05026827
Title: Iyengar Yoga as a Probe of Prolonged Grief Disorder Neurobiology
Brief Title: Iyengar Yoga for Prolonged Grief Disorder
Acronym: Yoga
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Joseph Goveas, Professor, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 00003864
Record Dates: First submitted 2021-08-24; First posted 2021-08-30 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Prolonged Grief Disorder
MeSH Terms: conditions — Prolonged Grief Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Iyengar Yoga (Experimental): Participants will engage in 10 weekly IY classes
  Interventions: Other: Iyengar Yoga
- Socialization Control (Active Comparator): Participants will engage in 10 weekly socialization control group sessions
  Interventions: Other: Socialization Control
- Healthy Comparison Group (No Intervention): A group of participants will also be followed for 10 weeks

INTERVENTIONS:
Other: Iyengar Yoga — Participation in Iyengar Yoga classes
  Arms: Iyengar Yoga
Other: Socialization Control — Participation in socialization control group sessions
  Arms: Socialization Control

SUMMARY:
Experiencing the death of a loved one is inevitable for older adults. Before the coronavirus disease 2019 (COVID-19) pandemic, over 2.5 million people died annually in the United States, including 52,000 in Wisconsin alone, and COVID-19 has added to this toll. Each person who dies leaves an average of five grieving people behind. Most grieving older adults are resilient and recover their pre-loss functioning within one year. However, in about 10%, acute grief becomes protracted and debilitating, leading to the development of prolonged grief disorder (PGD), a clinically diagnosable mental health condition. PGD in older adults increases the risk for poorer medical, mental health, and cognitive outcomes; lower quality of life; disability; premature mortality; and suicide. Despite the magnitude of this problem, the neurobiology of PGD in older adults is poorly understood. By using Iyengar Yoga (IY) as a probe for PGD neurobiology, this pilot project aims to address this critical gap.

DETAILED DESCRIPTION:
Our goal is to conduct a pilot study to examine in PGD the modulating effects of 10-week IY on circulating endocannabinoid and emotion processing brain circuit, and the associations between biological changes and clinical response.

ELIGIBILITY:
Inclusion Criteria:

* Male or female greater than or equal to 40 years of age
* Bereavement >6 months
* Score greater than or equal to 25 on the Inventory of Complicated Grief (ICG)
* Presence of PGD (subsyndromal and syndromal)
* Adequate visual and auditory acuity

Exclusion Criteria:

* Delirium/unstable medical conditions
* Lifetime history of neurological illnesses: seizures, stroke, dementia of any etiology, severe head injury, brain tumor or surgery
* Serious back, joint or neck injuries within the past 3 months
* Currently practicing yoga
* Gross structural abnormalities on T1-weighted images
* Lifetime history of the following psychiatric disorders: bipolar or psychotic disorders, including psychotic depression
* Current alcohol/drug abuse or dependence
* Magnetic resonance imaging (MRI) contraindications
* Acute suicidality

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2021-08-30 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in circulating endocannabinoid concentrations | 10 weeks
  Change in circulating endocannabinoids from baseline to post-intervention

SECONDARY OUTCOMES:
Change in neural activity measured using Functional magnetic resonance imaging (fMRI) | 10 weeks
  Change in neural activity from baseline to post-intervention
Inventory of Complicated Grief (ICG) scale score change | 10 weeks
  ICG score ranges from 0 to 76 (higher scores indicate worse outcome)

CONTACTS AND LOCATIONS:
Locations (1):
- Medical College of Wisconsin, Wauwatosa, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Goveas JS, Hwang G, McAuliffe TL, Blair NP, Webber A, Claesges SA, Murphy LM, Chandler K, Reynolds CF, Hainsworth KR. Iyengar yoga and health education interventions for prolonged grief disorder in later life: feasibility of a randomized controlled pilot trial. Sci Rep. 2025 Dec 24;15(1):44604. doi: 10.1038/s41598-025-28397-5. PMID 41444366